CLINICAL TRIAL: NCT04749173
Title: A Double-blind, Randomized, Placebo-controlled, Single-ascending Dose Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic Properties of Niclosamide Injectable (DWRX2003) Following Intramuscular Administration in Healthy Volunteers
Brief Title: To Assess the Safety, Tolerability and Pharmacokinetic Properties of Niclosamide Injectable (DWRX2003) Which is the Treatment of COVID-19 in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1516101
Record Dates: First submitted 2021-01-20; First posted 2021-02-11 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (96 mg) (Experimental): - Ventrogluteal area: 48 mg/0.2 mL x 2 sites
  Interventions: Drug: DWRX2003, 96mg
- Cohort 2 (432 mg) (Experimental): * Deltoid area: 72 mg/0.3 mL x 2 sites
  * Ventrogluteal area: 144 mg/0.6 mL x 2 sites
  Interventions: Drug: DWRX2003, 432mg
- Cohort A (144 mg) (Experimental): - Deltoid area: 72 mg/0.3 mL x 2 sites
  Interventions: Drug: DWRX2003, 144mg
- Cohort B (144 mg) (Experimental): - Ventrogluteal area: 72 mg/0.3 mL x 2 sites
  Interventions: Drug: DWRX2003, 144mg

INTERVENTIONS:
Drug: DWRX2003, 96mg — Drug: Placebo Intramuscularly injection at predefined injection sites
  Arms: Cohort 1 (96 mg)
Drug: DWRX2003, 432mg — Drug: Placebo Intramuscularly injection at predefined injection sites
  Arms: Cohort 2 (432 mg)
Drug: DWRX2003, 144mg — Drug: Placebo Intramuscularly injection at predefined injection sites
  Arms: Cohort A (144 mg)
Drug: DWRX2003, 144mg — Drug: Placebo Intramuscularly injection at predefined injection sites
  Arms: Cohort B (144 mg)

SUMMARY:
This Phase I study is a double-blind, randomized, placebo-controlled study designed to assess the safety, tolerability and PK profile of single intramuscular doses of DWRX2003 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 or older and 55 or younger at the time of screening test
2. A person who weighs 55.0 kg or more and whose BMI (body mass index) is above 18.0 and below 29.9;
3. A person who has listened to the detailed explanation of this clinical trial and fully understood, decided to participate voluntarily, and agreed in writing before the screening procedure.
4. A person who is eligible for this test when determining the person in charge of the test (or co-researcher who has been commissioned) due to physical examination, clinical laboratory examination, or examination.
5. A person who has been tested negative for Corona-19 virus (COVID-19) infection conducted during a screening visit.
6. A person who has agreed to use medically acceptable contraception during the pre-clinical trial period;

Exclusion Criteria:

1. A person with a history or medical condition that includes one or more of the following diseases:

   1. A person who is hypersensitive or has an history of overreaction to a clinical trial medication (or a component of a clinical trial medication) or emergency medication (epinephrine, dexamethasone, etc.)
   2. hepatitis B (active hepatitis B or carrier), hepatitis C, human immunodeficiency virus (HIV), or syphilis infection (unless fully cured in case of hepatitis B virus history)
   3. A person who is deemed clinically significant in determining the test manager (or a joint researcher) for the past or present history of asthma, rash, vascular edema, eczema, etc.
   4. A person who has clinical significance, liver, kidney, nervous system, respiratory system, endocrine system, blood, tumor, cardiovascular, urinary system, mental system disease, or history
   5. A person who has a history of malignant tumors in the past or present
   6. A person who has a history of whole-body anti-infection that has been terminated within 28 days prior to the administration of clinical trial medication, or a history of systemic or local infection that requires hospitalization or intravenous administration within 6 months before clinical trial medication is administered.
   7. A person who has undergone surgical intervention or surgery within 28 days prior to the administration of a clinical trial medication or is scheduled to undergo surgical procedures during the clinical trial period.
   8. A person who has a clinically significant blood clotting disorder or tendency to hemorrhagic
2. A person who shows the following results in a screening test:

   ﬁ A person whose blood level of AST (SGOT) and ALT (SGPT) exceeds twice the upper limit of the reference range ﬁ A person whose blood treatment line level exceeds the upper limit of the reference range or whose eGFR calculated by the Modification of Diet in Rental Disase (MDR) formula is less than 90ml/min/1.73㎡ ﬁ A person who has been found to be abnormal in the 12-lead ECG test ﬁ In the vital signs measured at the left position after a rest for more than three minutes, a person who showed a figure equivalent to systolic blood pressure of "90 mmHg or > 150 mmHg or extended blood pressure of "60 mmHg or >100 mmHg." ﬁ A person who has tested positive for serum (RPR Ab, anti-HIV (AIDS), HBs Ag, HCV Ab) ﬁ A person whose C-reactive protein (CRP) level is 1.5 times higher than the upper limit of the reference range.

   ﬁ In addition, a person who showed the results of a decision that the test manager (or a commissioned joint researcher) is clinically significant;
3. A person who has a history of drug abuse or has tested positive for abuse in urine drug testing
4. A person who participated in other clinical trials (including biological equivalence tests) within six months prior to the administration of the clinical trial medication (one test subject cannot participate in another cohort)
5. A person who has given full blood or blood donation within two months or within one month before the administration of a clinical trial medication or received blood transfusion within one month before the administration of a clinical trial medication.
6. A person who drinks continuously (21 units/week, 1 unit = 10 g of pure alcohol) within three months prior to administration of clinical trial medication, or cannot drink alcohol during hospitalization.
7. A person who smokes more than 10 cigarettes a day within one month prior to the administration of a clinical trial medication or who is not allowed to smoke during the hospitalization period.
8. A person who is not prohibited from eating anything other than food provided by the clinical testing institution during his/her admission period;
9. A male person who has a child plan or plans to donate sperm during the period prior to the clinical trial, or a female person who has a plan to conceive or breast-feed.
10. In addition to the above criteria, a person deemed inappropriate for the participation of a clinical trial by the person in charge of testing (or a joint researcher who has been delegated)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | follow-up 42 days after dosing
  Incidence, severity and causality of adverse events (AEs) and serious adverse events (SAEs) [ Time Frame: follow-up 42 days after dosing ]

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National university hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No